CLINICAL TRIAL: NCT01614977
Title: Comparison of Antibiotic Therapy Alone or Combined With Corticosteroids for the Treatment of Nontuberculous Mycobacterial Cervicofacial Lymphadenitis in Children: A Randomized Double-Blind Placebo-Controlled Study
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Technical problems.
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 6570
Record Dates: First submitted 2012-06-06; First posted 2012-06-08 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2011-08

CONDITIONS: Nontuberculous Mycobacterial Lymphadenitis.
Keywords: nontuberculous mycobacteria; corticosteroids; children; lymphadeniti; Therapeutic intervention in immunocompetent children with nontuberculous mycobacterial lymphadenitis.

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Methylprednisolone (Experimental): 1. Clarithromycin 15mg/Kg/day divided into 2 doses for 28 days.
  2. Rifambutin 20mg/Kg/day divided into 2 doses for 28 days.
  3. Methylprednisolone (Danalone) 1mg/Kg/dose twice daily for 14 days followed by 1mg/Kg/dose in the morning once daily for 14 days.
  Interventions: Drug: Methylprednisoline
- Placebo (No Intervention): 1. Clarithromycin 15mg/Kg/day divided into 2 doses for 28 days.
  2. Rifambutin 20mg/Kg/day divided into 2 doses for 28 days.
  3. placebo pills with an identical outward appearance and volume prescribed according to the same schedule.

INTERVENTIONS:
Drug: Methylprednisoline — Methylprednisolone (Danalone) 1mg/Kg/dose twice daily for 14 days followed by 1mg/Kg/dose in the morning once daily for 14 days,
  Arms: Methylprednisolone

SUMMARY:
Nontuberculous mycobacteriae (NTM) are a group of bacteria that typically cause infections of lymph nodes in the neck and face of otherwise healthy children.

There are currently 3 strategies to manage these infections. Yet, all are not "ideal" and each has downsides.

1. Surgery: removal of the affected lymph nodes is the most common approach but has the disadvantages of potential facial nerve paralysis, the possibility of recurrent infection that would require another operation and resolution with a cosmetically disturbing scar.
2. Antibiotics: The antibiotic courses are prolonged and are associated frequently with adverse reactions. It is unclear if this treatment has a significant effect on the "natural" resolution process of the infection.
3. Observation: follow-up the healing process without intervention. However the resolution may last a long period of time even more than a year. In almost all cases there will be spontaneous discharge of pus from the involved lymph nodes onto the skin that may last a few days. Later on a scar will form that may also be disturbing cosmetically.

The inflammatory response of the body to infections may occasionally be severe. As a matter of fact its harmful consequences can be sometimes more serious than those of the bacteria that cause the infection. Prednisone and other anti inflammatory drugs have properties that could possibly prevent this.

There is medical experience in using prednisone and similar drugs in addition to antibiotics in infectious diseases to decrease the inflammatory response against the infection. One of these infections is tuberculosis. The tuberculous bacteria have some common features with the nontuberculous mycobacteria. The investigators believe that the inflammatory process in infected lymph nodes with nontuberculous mycobacteria is the major cause for the discharge from the skin which later leads to the formation of a scar and to the prolonged resolution from the infection. Thus in order to hasten the resolution and to avoid formation of a neck or facial scar with its cosmetic consequences we suggest the use of prednisone in treating nontuberculus mycobacteria lymph nodes infections. Since prednisone depresses the inflammatory process as well as the immunity response, we chose to study the effect of prednisone combined with antibiotics (as the later will help to overcome the bacteria).

The purpose of the study is to determine whether the addition of prednisone to antibiotic treatment of nontuberculous mycobacteria lymph nodes infections in the neck and face of children can hasten the resolution process and improve its cosmetic results.

The diagnosis of nontuberculous mycobacteria lymph node infection will be based on evidence of bacterial growth in culture or on the presence of DNA of the bacteria in pus obtained from the involved lymph nodes by fine needle aspiration.

Generally healthy children with evidence of infection will be offered to participate in the study. They will be randomly assigned into the following 2 groups for 8 weeks treatment:

1. Antibiotics (2 types) and prednisone.
2. Antibiotics (2 types) and placebo (a material that tastes and look like prednisone but does not have any medical effect).

Prednisone will be given in a dose that will decrease into half twice: after 2 and after four weeks.

Follow-up visits for monitoring the inflammatory process and its resolution as well as adverse reactions will be done around 2 weeks, 4 weeks 3 months and 6-8 months after beginning therapy,

Blood tests and chest X-rays will be taken prior to the beginning of treatment. Blood tests will be also taken at the first follow-up visit.

A photo of the face neck and the site of the involved lymph nodes will be taken before starting therapy and at each of the follow-up visit.

DETAILED DESCRIPTION:
The objective of the study is to compare the effect of antimyocbacterial therapy alone or combined with corticosteroids for the treatment of NTM lymphadenitis in children.

The study will be conducted over a 3-year period in the Day Hospitalization Unit and ward C of the Schneider Children's Medical Center of Israel using a double- blind placebo-controlled design.

Eighty children aged 3 months to 20 years treated for laboratory-proven subacute/chronic NTM lymphadenitis at the Schneider Children's Medical Center of Israel will be enrolled in the study.

Children with any of the following findings will be excluded:

* congenital or acquired immunodeficiency
* chronic disease, such as diabetes mellitus, chronic renal failure, chronic liver disease, inflammatory bowel disease, or chronic arthritis
* immunosuppressive drug use (except inhaled steroids)
* elevated hepatocellular enzyme levels (more than twice the upper limit of normal) --- clinical suspicion of tuberculosis or a first-degree relative with tuberculosis.

ELIGIBILITY:
Inclusion Criteria:

* children aged 3 months to 20 years treated for laboratory-proven subacute/chronic NTM lymphadenitis.

Exclusion Criteria:

* congenital or acquired immunodeficiency
* chronic disease, such as diabetes mellitus, chronic renal failure, chronic liver disease, inflammatory bowel disease, or chronic arthritis
* immunosuppressive drug use (except inhaled steroids)
* elevated hepatocellular enzyme levels (more than twice the upper limit of normal)
* clinical suspicion of tuberculosis or a first-degree relative with tuberculosis.

Ages: 3 Months to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2011-10; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Resolution process of the involved lymph nodes | 3 years
  The primary end points of the study will be the color of the overlying skin, lymph node consistency, formulation of a fistula, and lesion area at the second and third follow-up visits.

SECONDARY OUTCOMES:
Adverse reaction to the medication | 3 years.
  The secondary end point will be any adverse reaction to the medication

CONTACTS AND LOCATIONS:
Overall Officials: Yishai Haimi Cohen, MD, Principal Investigator — SCMCI